CLINICAL TRIAL: NCT01090037
Title: TRK-100STP PhaseIIb/III Clinical Study - Chronic Renal Failure (Primary Glomerular Disease/Nephrosclerosis)
Brief Title: TRK-100STP Clinical Study - Chronic Renal Failure (Primary Glomerular Disease/Nephrosclerosis)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100CRS02/533-CL-003
Record Dates: First submitted 2010-03-08; First posted 2010-03-19 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Renal Failure; Glomerular Disease; Nephrosclerosis
Keywords: ESRD; Chronic Renal Failure; Prostaglandin; Prostacyclin; Asian Multinational Study
MeSH Terms: conditions — Kidney Failure, Chronic; Nephrosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRK-100STP (Experimental)
  Interventions: Drug: TRK-100STP high dose; Drug: TRK-100STP low dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRK-100STP high dose
  Arms: TRK-100STP
Drug: TRK-100STP low dose
  Arms: TRK-100STP
Drug: Placebo
  Arms: Placebo

SUMMARY:
In Chronic Renal Failure (CRF) patients with primary glomerular disease or nephrosclerosis as the primary disease:

* To confirm the superiority of TRK-100STP over placebo
* To determine the recommended therapeutic dose in the 2 doses of TRK-100STP
* To assess the safety of TRK-100STP

ELIGIBILITY:
Inclusion Criteria:

* The CRF patient with primary glomerular disease or nephrosclerosis as the primary disease
* The patient with progressive CRF

Exclusion Criteria:

* The patient with secondary glomerular disease
* The patient with CRF caused by pyelonephritis, interstitial/tubular nephritis, gouty kidney, polycystic kidney disease, or nephroureterolithiasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Renal composite endpoints [Time to first occurrence of one of the following events:] | 2-4 year
  (i) Doubling of SCr: Doubling of SCr is defined as a two-fold or greater increase in the SCr level, as compared with the baseline value
  (ii) ESRD (Occurrence of any of i-iii) i) Introduction of dialysis ii) Renal transplantation iii) Increase in SCr to 6.0 mg/dL or higher

CONTACTS AND LOCATIONS:
Locations (7):
- Beijing, China
- Hong Kong, Hong Kong
- Tokyo, Japan
- Kuala Lumpur, Malaysia
- Seoul, South Korea
- Taipei, Taiwan
- Bangkok, Thailand

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Nakamoto H, Fujita T, Origasa H, Isono M, Kurumatani H, Okada K, Kanoh H, Kiriyama T, Yamada S. A multinational phase IIb/III trial of beraprost sodium, an orally active prostacyclin analogue, in patients with primary glomerular disease or nephrosclerosis (CASSIOPEIR trial), rationale and study design. BMC Nephrol. 2014 Sep 19;15:153. doi: 10.1186/1471-2369-15-153. PMID 25233856